CLINICAL TRIAL: NCT02807623
Title: "Do NSAIDS or Executing Exercise Decrease Local Erythema, Site Swelling & Pain After INoculation: the NEED LESS PAIN Study"
Brief Title: Do NSAIDS or Executing Exercise Decrease Local Erythema, Site Swelling & Pain After INoculation
Acronym: NLP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Womack Army Medical Center (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 416446
Record Dates: First submitted 2016-06-10; First posted 2016-06-21 (Estimated); Results first posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Immune System and Related Disorders
MeSH Terms: interventions — Ibuprofen; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ibuprofen (Experimental): Randomized and double blinded study participants assigned to Group A intervention will receive an oral NSAID of ibuprofen 800 mgs three times a day for 48 hours.
  Interventions: Drug: Ibuprofen
- Placebo (Placebo Comparator): Randomized and double blinded study participants assigned to Group B intervention will receive an oral placebo three times a day for 48 hours starting immediately after influenza vaccine receipt.
  Interventions: Drug: oral placebo
- Compound Exercise of Push-ups (Experimental): Randomized study participants assigned to Group C will perform an exercise intervention of push-ups immediately after influenza vaccine receipt.
  Interventions: Behavioral: Compound Exercise of Push-ups

INTERVENTIONS:
Drug: Ibuprofen — The participants will take their first dose of the study drug immediately after influenza vaccine receipt. The medication will be blinded and dispensed by a research pharmacist. The participants will receive instructions on the dosing, frequency and a recommendation to take with food or milk and will be provided a snack with their first dose.
  Other Names: Motrin, Advil
  Arms: Ibuprofen
Behavioral: Compound Exercise of Push-ups — The participants will perform an exercise intervention of push-ups as immediately as possible but no more than 15 minutes after influenza vaccine receipt. The number of pushups performed will be at least 80% of the participants last Army Physical Fitness Test (APFT) score in one session. The number of pushups will be recorded. A baseline lactate fingerstick blood specimen will be collected with either the serology sample (if possible) or from the hand opposite the vaccine receipt arm prior to performing pushups and a second finger stick sample within 3-8 minutes, but no more than 15 minutes after vaccine receipt.
  Other Names: Push-ups
  Arms: Compound Exercise of Push-ups
Drug: oral placebo — The participants will take their first dose of the study drug immediately after influenza vaccine receipt. The medication will be blinded and dispensed by a research pharmacist. The participants will receive instructions on the dosing, frequency and a recommendation to take with food or milk and will be provided a snack with their first dose.
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this clinical investigation is to evaluate the efficacy and immunologic effects of a non-pharmacological exercise intervention (push-ups) compared to an oral NSAID (ibuprofen) and an oral placebo to decrease local injection site inflammation symptoms of delayed pain, erythema, and edema and any impact on serologic antibody immune response after influenza vaccine receipt.

DETAILED DESCRIPTION:
The study will evaluate the efficacy and immunologic effects of a non-pharmacological exercise intervention (push-ups) compared to an oral NSAID (ibuprofen) and a blinded oral placebo to decrease local injection site inflammation symptoms of delayed pain, erythema, and edema and any impact on serologic antibody immune response after influenza vaccine receipt. A healthy military cohort will be randomly assigned to either perform push-ups consistent with their army physical fitness score, or to take a blinded oral medication which will be an NSAID (ibuprofen) or an oral placebo. The study will require three visits for assessment: on the day of vaccine receipt, 48-72 hours later and 21 -28 days later. The assessment visits will include injection site inspection, an injection site photograph, completion of symptom diaries and a validated pain scale and a laboratory blood specimen at the first and third visit to measure antibody level changes. The exercise participants will also be required to provide 1-2 fingerstick blood samples to evaluate for lactate, which is a byproduct of anaerobic exercise to measure if level of exercise effort achieved anaerobic metabolism. The study will evaluate if either of the interventions impacted perceived delayed pain, physical signs of inflammation or antibody response as measured by serology.

ELIGIBILITY:
Inclusion Criteria:

Must:

1. Be Active Duty Service Members.
2. at least 18 years of age or older.
3. Be requiring and eligible for inactivated influenza vaccine receipt.
4. Be willing and able to complete the study protocol requirements.
5. Have a current Flu Screening Form with medical clearance to receive the influenza vaccination.

Exclusion Criteria:

Must Not:

1. Have already received influenza vaccine for the current season.
2. Have received any type of vaccine in the previous 72 hours.
3. Be on a medical profile resulting in current profile exemption from Physical Training of Upper 2 or Upper 3. (Upper extremity injury or illness)
4. Have preexisting symptoms of injury or infection or other local symptoms that would interfere with site assessment.
5. Be pregnant.
6. Have a history of allergy, intolerance, stomach bleeding or other medical exclusion for ibuprofen.
7. Have a history of stroke or coronary artery disease, such as uncontrolled high blood pressure or abnormal heart beat.
8. Has taken any topical or oral pain medications from the following medication classes in the past 24 hours prior to the start of the study: oral acetaminophen, opioids, tramadol, nonsteroidal anti-inflammatory drug (NSAID) or acetylsalicylic acid (ASA) or topical pain relievers or counterirritants of menthol, methyl salicylate, camphor menthols, and capsaicins.
9. Have any chronic or acute illness or treatment causing immunological suppression such as current oral steroid therapy, malignancy or chemotherapy or lung disease. (not including controlled asthma)
10. Currently participating in any other study

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-09; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurie A. Housel, MSN,FNP, Principal Investigator — Defense Health Agency Immunization Healthcare Branch
Locations (2):
- United States (2):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Womack Army Medical Center, Fort Bragg, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbott K, Fowler-Kerry S. The use of a topical refrigerant anesthetic to reduce injection pain in children. J Pain Symptom Manage. 1995 Nov;10(8):584-90. doi: 10.1016/0885-3924(95)00086-0. PMID 8594118
- [Background] Abuelkheir M, Alsourani D, Al-Eyadhy A, Temsah MH, Meo SA, Alzamil F. EMLA(R) cream: a pain-relieving strategy for childhood vaccination. J Int Med Res. 2014 Apr;42(2):329-36. doi: 10.1177/0300060513509473. Epub 2014 Feb 5. PMID 24501164
- [Background] Berberich FR, Landman Z. Reducing immunization discomfort in 4- to 6-year-old children: a randomized clinical trial. Pediatrics. 2009 Aug;124(2):e203-9. doi: 10.1542/peds.2007-3466. Epub 2009 Jul 13. PMID 19596729
- [Background] Bruunsgaard H, Hartkopp A, Mohr T, Konradsen H, Heron I, Mordhorst CH, Pedersen BK. In vivo cell-mediated immunity and vaccination response following prolonged, intense exercise. Med Sci Sports Exerc. 1997 Sep;29(9):1176-81. doi: 10.1097/00005768-199709000-00009. PMID 9309628
- [Background] Campbell JP, Edwards KM, Ring C, Drayson MT, Bosch JA, Inskip A, Long JE, Pulsford D, Burns VE. The effects of vaccine timing on the efficacy of an acute eccentric exercise intervention on the immune response to an influenza vaccine in young adults. Brain Behav Immun. 2010 Feb;24(2):236-42. doi: 10.1016/j.bbi.2009.10.001. Epub 2009 Oct 8. PMID 19818846
- [Background] Chambers CT, Taddio A, Uman LS, McMurtry CM; HELPinKIDS Team. Psychological interventions for reducing pain and distress during routine childhood immunizations: a systematic review. Clin Ther. 2009;31 Suppl 2:S77-S103. doi: 10.1016/j.clinthera.2009.07.023. PMID 19781437
- [Background] Cobb JE, Cohen LL. A randomized controlled trial of the ShotBlocker for children's immunization distress. Clin J Pain. 2009 Nov-Dec;25(9):790-6. doi: 10.1097/AJP.0b013e3181af1324. PMID 19851160
- [Background] Cohen Reis E, Holubkov R. Vapocoolant spray is equally effective as EMLA cream in reducing immunization pain in school-aged children. Pediatrics. 1997 Dec;100(6):E5. doi: 10.1542/peds.100.6.e5. PMID 9374583
- [Background] Das RR, Panigrahi I, Naik SS. The effect of prophylactic antipyretic administration on post-vaccination adverse reactions and antibody response in children: a systematic review. PLoS One. 2014 Sep 2;9(9):e106629. doi: 10.1371/journal.pone.0106629. eCollection 2014. PMID 25180516
- [Background] Dilli D, Kucuk IG, Dallar Y. Interventions to reduce pain during vaccination in infancy. J Pediatr. 2009 Mar;154(3):385-90. doi: 10.1016/j.jpeds.2008.08.037. Epub 2008 Oct 11. PMID 18849052
- [Background] Doedee AM, Boland GJ, Pennings JL, de Klerk A, Berbers GA, van der Klis FR, de Melker HE, van Loveren H, Janssen R. Effects of prophylactic and therapeutic paracetamol treatment during vaccination on hepatitis B antibody levels in adults: two open-label, randomized controlled trials. PLoS One. 2014 Jun 4;9(6):e98175. doi: 10.1371/journal.pone.0098175. eCollection 2014. PMID 24897504
- [Background] Gidudu JF, Walco GA, Taddio A, Zempsky WT, Halperin SA, Calugar A, Gibbs NA, Hennig R, Jovancevic M, Netterlid E, O'Connor T, Oleske JM, Varricchio F, Tsai TF, Seifert H, Schuind AE; Brighton Immunization Site Pain Working Group. Immunization site pain: case definition and guidelines for collection, analysis, and presentation of immunization safety data. Vaccine. 2012 Jun 22;30(30):4558-77. doi: 10.1016/j.vaccine.2012.03.085. Epub 2012 Apr 18. No abstract available. PMID 22521267
- [Background] Gidudu J, Kohl KS, Halperin S, Hammer SJ, Heath PT, Hennig R, Hoet B, Rothstein E, Schuind A, Varricchio F, Walop W; Brighton Collaboration Local Reactions Working Group for a Local Reaction at or near Injection Site. A local reaction at or near injection site: case definition and guidelines for collection, analysis, and presentation of immunization safety data. Vaccine. 2008 Dec 9;26(52):6800-13. doi: 10.1016/j.vaccine.2008.10.006. Epub 2008 Oct 23. PMID 18950670
- [Background] Edwards KM, Booy R. Effects of exercise on vaccine-induced immune responses. Hum Vaccin Immunother. 2013 Apr;9(4):907-10. doi: 10.4161/hv.23365. Epub 2013 Jan 14. PMID 23319202
- [Background] Edwards KM, Burns VE, Adkins AE, Carroll D, Drayson M, Ring C. Meningococcal A vaccination response is enhanced by acute stress in men. Psychosom Med. 2008 Feb;70(2):147-51. doi: 10.1097/PSY.0b013e318164232e. Epub 2008 Feb 6. PMID 18256346
- [Background] Edwards KM, Burns VE, Allen LM, McPhee JS, Bosch JA, Carroll D, Drayson M, Ring C. Eccentric exercise as an adjuvant to influenza vaccination in humans. Brain Behav Immun. 2007 Feb;21(2):209-17. doi: 10.1016/j.bbi.2006.04.158. Epub 2006 Jul 7. PMID 16824730
- [Background] Edwards KM, Burns VE, Reynolds T, Carroll D, Drayson M, Ring C. Acute stress exposure prior to influenza vaccination enhances antibody response in women. Brain Behav Immun. 2006 Mar;20(2):159-68. doi: 10.1016/j.bbi.2005.07.001. Epub 2005 Aug 15. PMID 16102936
- [Background] Edwards KM, Campbell JP, Ring C, Drayson MT, Bosch JA, Downes C, Long JE, Lumb JA, Merry A, Paine NJ, Burns VE. Exercise intensity does not influence the efficacy of eccentric exercise as a behavioural adjuvant to vaccination. Brain Behav Immun. 2010 May;24(4):623-30. doi: 10.1016/j.bbi.2010.01.009. Epub 2010 Jan 25. PMID 20102734
- [Background] Edwards KM, Pung MA, Tomfohr LM, Ziegler MG, Campbell JP, Drayson MT, Mills PJ. Acute exercise enhancement of pneumococcal vaccination response: a randomised controlled trial of weaker and stronger immune response. Vaccine. 2012 Oct 5;30(45):6389-95. doi: 10.1016/j.vaccine.2012.08.022. Epub 2012 Aug 22. PMID 22921739
- [Background] Gleeson M, Pyne DB, McDonald WA, Clancy RL, Cripps AW, Horn PL, Fricker PA. Pneumococcal antibody responses in elite swimmers. Clin Exp Immunol. 1996 Aug;105(2):238-44. doi: 10.1046/j.1365-2249.1996.d01-752.x. PMID 8706328
- [Background] Taddio A, Lord A, Hogan ME, Kikuta A, Yiu A, Darra E, Bruinse B, Keogh T, Stephens D. A randomized controlled trial of analgesia during vaccination in adults. Vaccine. 2010 Jul 19;28(32):5365-9. doi: 10.1016/j.vaccine.2010.05.015. Epub 2010 May 16. PMID 20483194
- [Background] Hogan ME, Kikuta A, Taddio A. A systematic review of measures for reducing injection pain during adult immunization. Vaccine. 2010 Feb 10;28(6):1514-21. doi: 10.1016/j.vaccine.2009.11.065. Epub 2009 Dec 8. PMID 20003927
- [Background] Irwin MR, Olmstead R, Oxman MN. Augmenting immune responses to varicella zoster virus in older adults: a randomized, controlled trial of Tai Chi. J Am Geriatr Soc. 2007 Apr;55(4):511-7. doi: 10.1111/j.1532-5415.2007.01109.x. PMID 17397428
- [Background] Jackson LA, Dunstan M, Starkovich P, Dunn J, Yu O, Nelson JC, Rees T, Zavitkovsky A. Prophylaxis with acetaminophen or ibuprofen for prevention of local reactions to the fifth diphtheria-tetanus toxoids-acellular pertussis vaccination: a randomized, controlled trial. Pediatrics. 2006 Mar;117(3):620-5. doi: 10.1542/peds.2005-1217. PMID 16510639
- [Background] Keylock KT, Lowder T, Leifheit KA, Cook M, Mariani RA, Ross K, Kim K, Chapman-Novakofski K, McAuley E, Woods JA. Higher antibody, but not cell-mediated, responses to vaccination in high physically fit elderly. J Appl Physiol (1985). 2007 Mar;102(3):1090-8. doi: 10.1152/japplphysiol.00790.2006. Epub 2006 Nov 9. PMID 17095638
- [Background] Kohl KS, Walop W, Gidudu J, Ball L, Halperin S, Hammer SJ, Heath P, Hennig R, Rothstein E, Schuind A, Varricchio F; Brighton Collaboration Local Reactions Working Group for Induration at or near Injection Site. Induration at or near injection site: case definition and guidelines for collection, analysis, and presentation of immunization safety data. Vaccine. 2007 Aug 1;25(31):5839-57. doi: 10.1016/j.vaccine.2007.04.062. Epub 2007 May 8. No abstract available. PMID 17553602
- [Background] Kohl KS, Walop W, Gidudu J, Ball L, Halperin S, Hammer SJ, Heath P, Varricchio F, Rothstein E, Schuind A, Hennig R; Brighton Collaboration Local Reaction Working Group for Swelling at or near Injection Site. Swelling at or near injection site: case definition and guidelines for collection, analysis and presentation of immunization safety data. Vaccine. 2007 Aug 1;25(31):5858-74. doi: 10.1016/j.vaccine.2007.04.056. Epub 2007 May 11. No abstract available. PMID 17548132
- [Background] Kohut ML, Arntson BA, Lee W, Rozeboom K, Yoon KJ, Cunnick JE, McElhaney J. Moderate exercise improves antibody response to influenza immunization in older adults. Vaccine. 2004 Jun 2;22(17-18):2298-306. doi: 10.1016/j.vaccine.2003.11.023. PMID 15149789
- [Background] Kohut ML, Cooper MM, Nickolaus MS, Russell DR, Cunnick JE. Exercise and psychosocial factors modulate immunity to influenza vaccine in elderly individuals. J Gerontol A Biol Sci Med Sci. 2002 Sep;57(9):M557-62. doi: 10.1093/gerona/57.9.m557. PMID 12196490
- [Background] Kristjansdottir O, Kristjansdottir G. Randomized clinical trial of musical distraction with and without headphones for adolescents' immunization pain. Scand J Caring Sci. 2011 Mar;25(1):19-26. doi: 10.1111/j.1471-6712.2010.00784.x. PMID 20409050
- [Background] Long JE, Ring C, Bosch JA, Eves F, Drayson MT, Calver R, Say V, Allen D, Burns VE. A life-style physical activity intervention and the antibody response to pneumococcal vaccination in women. Psychosom Med. 2013 Oct;75(8):774-82. doi: 10.1097/PSY.0b013e3182a0b664. Epub 2013 Aug 6. PMID 23922400
- [Background] Long JE, Ring C, Drayson M, Bosch J, Campbell JP, Bhabra J, Browne D, Dawson J, Harding S, Lau J, Burns VE. Vaccination response following aerobic exercise: can a brisk walk enhance antibody response to pneumococcal and influenza vaccinations? Brain Behav Immun. 2012 May;26(4):680-7. doi: 10.1016/j.bbi.2012.02.004. Epub 2012 Feb 22. PMID 22386744
- [Background] Maiden MJ, Benton GN, Bourne RA. Effect of warming adult diphtheria-tetanus vaccine on discomfort after injection: a randomised controlled trial. Med J Aust. 2003 May 5;178(9):433-6. doi: 10.5694/j.1326-5377.2003.tb05284.x. PMID 12720508
- [Background] Manley J, Taddio A. Acetaminophen and ibuprofen for prevention of adverse reactions associated with childhood immunization. Ann Pharmacother. 2007 Jul;41(7):1227-32. doi: 10.1345/aph.1H647. Epub 2007 May 22. PMID 17519301
- [Background] Mawhorter S, Daugherty L, Ford A, Hughes R, Metzger D, Easley K. Topical vapocoolant quickly and effectively reduces vaccine-associated pain: results of a randomized, single-blinded, placebo-controlled study. J Travel Med. 2004 Sep-Oct;11(5):267-72. doi: 10.2310/7060.2004.19101. PMID 15544709
- [Background] Nakashima Y, Harada M, Okayama M, Kajii E. Analgesia for pain during subcutaneous injection: effectiveness of manual pressure application before injection. Int J Gen Med. 2013 Sep 25;6:817-20. doi: 10.2147/IJGM.S50125. eCollection 2013. PMID 24101880
- [Background] Nilsson S, Forsner M, Finnstrom B, Morelius E. Relaxation and guided imagery do not reduce stress, pain and unpleasantness for 11- to 12-year-old girls during vaccinations. Acta Paediatr. 2015 Jul;104(7):724-9. doi: 10.1111/apa.13000. Epub 2015 Apr 22. PMID 25762426
- [Background] Pascoe AR, Fiatarone Singh MA, Edwards KM. The effects of exercise on vaccination responses: a review of chronic and acute exercise interventions in humans. Brain Behav Immun. 2014 Jul;39:33-41. doi: 10.1016/j.bbi.2013.10.003. Epub 2013 Oct 11. PMID 24126151
- [Background] Porter CK, Bowens MJ, Tribble DR, Putnam SD, Sanders JW, Riddle MS. Attitudes towards vaccines and infectious disease risk among U.S. troops. Hum Vaccin. 2008 Jul-Aug;4(4):298-304. doi: 10.4161/hv.4.4.5802. Epub 2008 Feb 27. No abstract available. PMID 18398299
- [Background] Prymula R, Siegrist CA, Chlibek R, Zemlickova H, Vackova M, Smetana J, Lommel P, Kaliskova E, Borys D, Schuerman L. Effect of prophylactic paracetamol administration at time of vaccination on febrile reactions and antibody responses in children: two open-label, randomised controlled trials. Lancet. 2009 Oct 17;374(9698):1339-50. doi: 10.1016/S0140-6736(09)61208-3. PMID 19837254
- [Background] Ranadive SM, Cook M, Kappus RM, Yan H, Lane AD, Woods JA, Wilund KR, Iwamoto G, Vanar V, Tandon R, Fernhall B. Effect of acute aerobic exercise on vaccine efficacy in older adults. Med Sci Sports Exerc. 2014 Mar;46(3):455-61. doi: 10.1249/MSS.0b013e3182a75ff2. PMID 23924918
- [Background] Rose MA, Juergens C, Schmoele-Thoma B, Gruber WC, Baker S, Zielen S. An open-label randomized clinical trial of prophylactic paracetamol coadministered with 7-valent pneumococcal conjugate vaccine and hexavalent diphtheria toxoid, tetanus toxoid, 3-component acellular pertussis, hepatitis B, inactivated poliovirus, and Haemophilus influenzae type b vaccine. BMC Pediatr. 2013 Jun 21;13:98. doi: 10.1186/1471-2431-13-98. PMID 23786774
- [Background] Russell K, Nicholson R, Naidu R. Reducing the pain of intramuscular benzathine penicillin injections in the rheumatic fever population of Counties Manukau District Health Board. J Paediatr Child Health. 2014 Feb;50(2):112-7. doi: 10.1111/jpc.12400. Epub 2013 Oct 18. PMID 24134180
- [Background] Shah V, Taddio A, Rieder MJ; HELPinKIDS Team. Effectiveness and tolerability of pharmacologic and combined interventions for reducing injection pain during routine childhood immunizations: systematic review and meta-analyses. Clin Ther. 2009;31 Suppl 2:S104-51. doi: 10.1016/j.clinthera.2009.08.001. PMID 19781433
- [Background] Schuler PB, Leblanc PA, Marzilli TS. Effect of physical activity on the production of specific antibody in response to the 1998-99 influenza virus vaccine in older adults. J Sports Med Phys Fitness. 2003 Sep;43(3):404. PMID 14625524
- [Background] Sparks L. Taking the "ouch" out of injections for children. Using distraction to decrease pain. MCN Am J Matern Child Nurs. 2001 Mar-Apr;26(2):72-8. doi: 10.1097/00005721-200103000-00005. PMID 11265439
- [Background] Taddio A, Appleton M, Bortolussi R, Chambers C, Dubey V, Halperin S, Hanrahan A, Ipp M, Lockett D, MacDonald N, Midmer D, Mousmanis P, Palda V, Pielak K, Riddell RP, Rieder M, Scott J, Shah V. Reducing the pain of childhood vaccination: an evidence-based clinical practice guideline (summary). CMAJ. 2010 Dec 14;182(18):1989-95. doi: 10.1503/cmaj.092048. Epub 2010 Nov 22. No abstract available. PMID 21098067
- [Background] Taddio A, Chambers CT, Halperin SA, Ipp M, Lockett D, Rieder MJ, Shah V. Inadequate pain management during routine childhood immunizations: the nerve of it. Clin Ther. 2009;31 Suppl 2:S152-67. doi: 10.1016/j.clinthera.2009.07.022. PMID 19781434
- [Background] Taddio A, Ilersich AL, Ipp M, Kikuta A, Shah V; HELPinKIDS Team. Physical interventions and injection techniques for reducing injection pain during routine childhood immunizations: systematic review of randomized controlled trials and quasi-randomized controlled trials. Clin Ther. 2009;31 Suppl 2:S48-76. doi: 10.1016/j.clinthera.2009.07.024. PMID 19781436
- [Background] Woods JA, Keylock KT, Lowder T, Vieira VJ, Zelkovich W, Dumich S, Colantuano K, Lyons K, Leifheit K, Cook M, Chapman-Novakofski K, McAuley E. Cardiovascular exercise training extends influenza vaccine seroprotection in sedentary older adults: the immune function intervention trial. J Am Geriatr Soc. 2009 Dec;57(12):2183-91. doi: 10.1111/j.1532-5415.2009.02563.x. PMID 20121985
- [Background] Yalcin SS, Gumus A, Yurdakok K. Prophylactic use of acetaminophen in children vaccinated with diphtheria-tetanus-pertussis. World J Pediatr. 2008 May;4(2):127-9. doi: 10.1007/s12519-008-0025-7. PMID 18661769
- [Background] Afluria US Package Insert for 2015-2016. 2015. bioCSL version 44. Retrieved from http://www.fda.gov/downloads/BiologicsBloodVaccines/Vaccines/ApprovedProducts/UCM263239.pdf
- [Background] Defense Health Agency (2004). Clinical guidelines for managing adverse events after vaccination. Defense Health Agency Immunization Health Care Branch. US Army Medical Command, Falls Church, VA.
- [Background] Díez-Domingo, J., Planelles, M., Baldó, J., Ballester, A., Núñez, F., Jubert, A., & Dominguez-Granados, R. (1998). Ibuprofen prophylaxis for adverse reactions to diphtheria-tetanus-pertussis vaccination: a randomized trial. Current Therapeutic Research, 59(8), 579-588.
- [Background] Fluarix US Package Insert. 2014. GlaxoSmithKline.
- [Background] Fluzone US Package Insert. June 2014. Sanofi Pasteur, Inc.
- [Background] Flublock US Package Insert. October 2014. Protein Sciences Corporation
- [Background] Flucelvax US Package Insert. March 2014. Novartis Vaccines and Diagnostics, Inc.
- [Background] Flulavel US Package Insert. May 2014. GlaxoSmithKline.
- [Background] Fluvirin US Package Insert. April 2014. Novartis Vaccines and Diagnostics, Inc.
- [Background] Hayat, H., Khan, Parwez S. & Hayat, G. (2011). The effect of prophylactic paracetamol administration on adverse reactions following DTP vaccination. Eastern Journal of Medicine 16, 258-260.
- [Background] Schuler PB, Lloyd LK, Leblanc PA, Clapp TA, Abadie BR, Collins RK. The effect of physical activity and fitness on specific antibody production in college students. J Sports Med Phys Fitness. 1999 Sep;39(3):233-9. PMID 10573666
- [Background] Whitham M, Blannin AK. The effect of exercise training on the kinetics of the antibody response to influenza vaccination. J Sports Sci. 2003 Dec;21(12):991-1000. doi: 10.1080/0264041031000140464. PMID 14748456

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 315 active-duty US Military Service Members due to receive injectable influenza vaccine (IIV) were recruited via flyers or verbal briefing from the Fort Bragg, North Carolina 82'nd Airborne Soldier Readiness Center and Walter Reed National Military Medical Center between 9/19/2016 and 11/6/2018.
Pre-assignment Details: Of these 315 subjects, 15 were excluded due to the following reasons: 4 did not meet inclusion criteria, 2 declined to participate, and 9 are identified as other reasons. 300 were randomized to 1 of 3 arms. However, only 233 of the 300 returned for follow-up visits. Thus results are based on data from those 233 participants with completed data.
Period: Overall Study
Arm/Group | Ibuprofen | Placebo | Compound Exercise of Push-ups
Started | 98 | 100 | 102
Completed | 75 | 79 | 79
Not Completed | 23 | 21 | 23
Not completed — Lost to Follow-up | 23 | 18 | 22
Not completed — Drug intolerance | 0 | 1 | 0
Not completed — incomplete blood draw | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen | Placebo | Compound Exercise of Push-ups | Total
Number analyzed (Participants) | 75 | 81 | 77 | 233
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 75 | 81 | 77 | 233
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.13 (6.119) | 25.33 (5.239) | 25.95 (5.426) | 25.79 (5.583)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 11 | 38
  Male | 64 | 65 | 66 | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 61 | 53 | 162
  Not Hispanic or Latino | 18 | 18 | 17 | 53
  Unknown or Not Reported | 9 | 2 | 7 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 22 | 13 | 45
  White | 38 | 39 | 40 | 117
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 27 | 20 | 24 | 71
Region of Enrollment [Number; unit: participants]
  United States | 75 | 81 | 77 | 233

OUTCOME MEASURES:

1. Primary Outcome: Level of Pain
Description: Level of Pain will be measured by validated pain scale, using a scale of 0 ( best, no pain) to 10 (worst, as bad as imaginable, completely interferes).
Time Frame: baseline, 48-72 hours and at 21-28 days ( 3 points )
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ibuprofen | Placebo | Compound Exercise of Push-ups
Number analyzed (Participants) | 75 | 80 | 78
units on a scale
  Visit 1 | .39 (1.384) | .19 (.713) | .14 (.639)
  Visit 2 | .56 (1.626) | .22 (.741) | .19 (.650)
  Visit 3 | .28 (1.122) | .06 (0.401) | .13 (.745)

2. Secondary Outcome: Serologic Response - A/California/7/2009
Description: Baseline lab specimen (visit 1, day 0, before immunization) and repeated between 21-28 days (visit 3) after immunization to measure serologic response
Time Frame: Day 0 and between 21-28 days (2 points)
Measure: Mean (Standard Deviation); unit: Titer
Arm/Group | Placebo | Ibuprofen | Compound Exercise of Push-ups
Number analyzed (Participants) | 32 | 32 | 45
Titer
  Baseline (day 0, visit 1) | 216.75 (182.072) | 171.00 (105.970) | 214.80 (171.742)
  Followup (between 21-28 days, visit 3) | 343.03 (216.797) | 239.25 (120.223) | 345.09 (217.495)

3. Secondary Outcome: Serologic Response - A/Hong Kong / 4801/2014
Description: as for outcome 2
Time Frame: Day 0 and between 21-28 days (2 points)
Measure: Mean (Standard Deviation); unit: Titer
Arm/Group | Placebo | Ibuprofen | Compound Exercise of Push-ups
Number analyzed (Participants) | 32 | 32 | 45
Titer
  Baseline (day 0, visit 1) | 221.09 (263.64) | 177.78 (165.489) | 149.22 (146.387)
  Followup (between 21-28 days, visit 3) | 296.66 (299.001) | 243.13 (203.461) | 232.58 (176.394)

4. Secondary Outcome: Serologic Response - B/Phuket/3073/2013
Description: as for outcome 2
Time Frame: Day 0 and between 21-28 days (2 points)
Measure: Mean (Standard Deviation); unit: Titer
Arm/Group | Placebo | Ibuprofen | Compound Exercise of Push-ups
Number analyzed (Participants) | 32 | 32 | 45
Titer
  Baseline (day 0, visit 1) | 36.69 (44.586) | 40.16 (60.321) | 32.89 (33.857)
  Followup (between 21-28 days, visit 3) | 44.78 (43.773) | 47.34 (58.976) | 49.07 (39.578)

5. Secondary Outcome: Serologic Response - B/Brisbane/60/2008
Description: as for outcome 2
Time Frame: Day 0 and between 21-28 days (2 points)
Measure: Mean (Standard Deviation); unit: Titer
Arm/Group | Placebo | Ibuprofen | Compound Exercise of Push-ups
Number analyzed (Participants) | 32 | 32 | 45
Titer
  Baseline (day 0, visit 1) | 26.09 (31.308) | 17.41 (12.271) | 26.00 (35.833)
  Followup (between 21-28 days, visit 3) | 34.09 (29.977) | 25.47 (18.30) | 41.02 (39.199)

6. Secondary Outcome: Participants With Erythema
Description: Reddening of the skin at vaccination site reported as the total number of participants with erythema over the duration of the study.
Time Frame: baseline, 48- 72 hours, 21-28 days (3 points)
Population: Statistical analysis of participants with erythema post-vaccination was not performed due to no cases of erythema reported by participants or observed by research staff.
Measure: Count of Participants; unit: Participants
Groups:
- Baseline: Participants were evaluated for reddening of the skin at the vaccination site immediately after influenza vaccine receipt.
- 48-72 Hours After Vaccination: Participants were evaluated for reddening of the skin at the vaccination site 48-72 hours after influenza vaccine receipt.
- 21-28 Days After Vaccination: Participants were evaluated for reddening of the skin at the vaccination site 21-28 days after influenza vaccine receipt.
Arm/Group | Baseline | 48-72 Hours After Vaccination | 21-28 Days After Vaccination
Number analyzed (Participants) | 233 | 233 | 233
Participants | 0 | 0 | 0

7. Secondary Outcome: Participants With Edema
Description: Swelling at vaccination site
Time Frame: baseline, 48-72 hours, and 21- 28 days (3 points)
Population: Statistical analysis of participants with edema post-vaccination was not performed due to no cases of edema reported by participants or observed by research staff.
Measure: Count of Participants; unit: Participants
Groups:
- Baseline: Participants were evaluated for swelling at the vaccination site immediately after influenza vaccine receipt.
- 48-72 Hours After Vaccination: Participants were evaluated for swelling at the vaccination site 48-72 hours after influenza vaccine receipt.
- 21-28 Days After Vaccination: Participants were evaluated for swelling at the vaccination site 21-28 days after influenza vaccine receipt.
Arm/Group | Baseline | 48-72 Hours After Vaccination | 21-28 Days After Vaccination
Number analyzed (Participants) | 233 | 233 | 233
Participants | 0 | 0 | 0

8. Other Pre Specified Outcome: Lactate
Description: A Lactate meter was used to test the exercise group for lactate readings. Two lactate tests was performed for the exercise group at Visit 1, both pre and post Influenza vaccination. The first lactate reading was taken after the blood draw.The second lactate reading was obtained from a fingerstick from the hand opposite to the vaccination arm, ideally within 3-8 minutes after the study subject completes pushups.
Time Frame: Immediately prior to Influenza vaccine and 3-8 minutes after Influenza vaccine was administered and after push-ups were completed.
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Compound Exercise of Push-ups
Number analyzed (Participants) | 77
mmol/L
  Lactate before pushups | 1.51 [1.27 to 1.75]
  Lactate after pushups | 7.69 [7.11 to 8.27]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each study participant beginning the day of enrollment and throughout the completion of the study at visit three day 21-28.
Arm/Group | Ibuprofen | Placebo | Compound Exercise of Push-ups
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/100 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/100 | 0/102
Other Adverse Events (participants affected / at risk) | 0/98 | 1/100 | 0/102
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibuprofen (N=98) | Placebo (N=100) | Compound Exercise of Push-ups (N=102)
dysmenhorrhea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) — Subject c/o lower abdominal pain after taking drug dose #3; seen clinically. Subject was unblinded and determined to have taken placebo and not study related, other than didn't take usual ibuprofen for menstrual cramps due to study participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT02807623/Prot_SAP_000.pdf